CLINICAL TRIAL: NCT03444831
Title: Buspirone Plus Omeprazole for Functional Dyspepsia: A Randomised Placebo Clinical Trial
Brief Title: Buspirone Plus Omeprazole for Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Meisam AbdarEsfahani, Mediacal Doctor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 166681
Record Dates: First submitted 2018-02-10; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Buspirone; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone plus Omeprazole (Experimental)
  Interventions: Drug: Buspirone
- Placebo plus Omeprazole (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Buspirone — Buspirone 5mg used QID a day after meal plus 20mg omeprazole before breakfast.
  Other Names: Omeprazole
  Arms: Buspirone plus Omeprazole
Drug: Placebo Oral Tablet — Buspirone placebo QID after meal plus 20mg omeprazole before breakfast.
  Other Names: omeprazole
  Arms: Placebo plus Omeprazole

SUMMARY:
This study is a double-blinded Randomised clinical trial aim to compare buspirone plus omeprazole with placebo plus omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* being over 18-year-old, Rome III criteria for FD
* normal upper endoscopy within five years
* negative Urease test for H-pylori
* acceptance informed concept form.

Exclusion Criteria:

* denied to get these medications
* taking other drugs for FD
* patients with the organic gastrointestinal disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
70 patients With functional dyspepsia symptoms, Change From Baseline by asking about symptoms at 4 Weeks after using buspirone or placebo | 4 weeks taking buspirone plus omeprasole or taking placebo plus omeprasloe
  Global symptom measured through a checklist of dyspepsia symptoms at first visit and four weeks after

IPD SHARING:
Plan to Share IPD: Undecided